CLINICAL TRIAL: NCT00006331
Title: Prospective Controlled Study of Posttransplant Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00042-1699; M01RR000042 (NIH)
Record Dates: First submitted 2000-10-04; First posted 2000-10-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Diabetes Mellitus; Kidney Failure
Keywords: Kidney transplantation; Immunology
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency | interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: renal transplant

SUMMARY:
Research participants will be asked to undergo complete medical history, physical examination and blood tests. The purpose of these tests is to determine whether persons are predisposed to develop diabetes mellitus after kidney transplantation and also to make an early diagnosis if a patient develops diabetes mellitus. Medical information collected as part of the standard transplant evaluation and posttransplant medical care may be incorporated into this study. It is important to realize that research subjects will not be given an experimental drug as part of this study.

After kidney transplantation, research subjects will be followed in the posttransplant clinic visits. The study will last up to 6 months. During this time the subjects may be asked to participate in clinical assessment visits (medical history and physical examination), and also during the third or fourth month after transplant will be asked to do a repeat glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Fasting Plasma Glucose (FPG) <126mg/dl.
* No history of diabetes mellitus or treatment with oral antidiabetic agent or insulin.
* ESRD or chronic renal failure with CrCl <= 20cc/min per 1.73m2.
* Waiting list registration for cadaveric or set date for living donor renal transplantation.
* Willingness and ability to understand and give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- 3914 Taubman Center, Ann Arbor, Michigan, United States